CLINICAL TRIAL: NCT03428893
Title: MyTherEx: Mobile Technology to Support Physical Therapist Directed Exercise for People Aging With Arthritis
Brief Title: Mobile Technology to Support Physical Therapy Exercise
Acronym: MyTherEx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Nancy Gell, Assistant Professor, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17_0663
Record Dates: First submitted 2018-02-05; First posted 2018-02-12 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Osteoarthritis of Knee; Osteoarthritis Of Hip
Keywords: Exercise, mhealth, physical therapy
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Application Group (Experimental): The mobile app group will receive physical therapy as determined by the physical therapist and agree to receive the home exercise prescription using a mobile app on their phone or personal tablet
  Interventions: Device: Mobile Application
- Control (No Intervention): The control group will receive physical therapy as determined by the physical therapist based on clinical practice guidelines and will receive the home exercise program in the traditional way through paper exercise handouts

INTERVENTIONS:
Device: Mobile Application — Participants will receive usual care physical therapy guided by Clinical Practice Guidelines and based on individual symptoms and need over 7 in-person visits. Measures will be collected by the physical therapist related to leg strength, balance, fitness, and mobility as part of the usual care physical therapy evaluation and follow-up. The treating physical therapist will negotiate the physical therapy intervention based on patient preferences and goals and assessment findings. Using clinical practice guidelines, the intervention for the research participants is expected to address deficits in strength, mobility, balance, and cardiovascular endurance. Exercise prescription will be provided using the Wellpepper physical therapy exercise prescription mobile app.
  Arms: Mobile Application Group

SUMMARY:
Osteoarthritis is the leading cause of disability in the U.S, particularly in older adults. Exercise is an evidence-based treatment option that improves pain and disability outcomes in adults with osteoarthritis, but adherence to prescribed exercise is generally low. Technology such as mobile applications (apps) for smartphones and tablets offers the potential to support exercise adherence through evidence-based components and enhanced communication between physical therapists and patients. The investigators aim to test mobile app-supported physical therapy exercise prescription compared to standard care. The investigators propose to use a two-arm randomized control trial with subjects in the intervention receiving mobile app-supported physical therapy exercise prescription and the control group receiving usual care physical therapy exercise prescription (paper handouts and verbal instruction). No known studies have assessed the impact of technological integration on adherence with PT exercises for OA. Current approaches such as therapist drawn pictures, hand-written or print-ready instructions do not account for patient communication preferences or ability to translate drawings into physical action. Mobile technology offers a potential solution to patient-centered care but has not been evaluated. This study will provide valuable information on effectiveness and user perspectives to key stakeholders such as patients, health care administrators, physical therapists and app designers.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the leading cause of disability in the U.S. The rate of activity limitation due to OA is progressing faster than expected while prevalence is projected to increase as a result of the obesity epidemic and population aging, making it a major public health problem. Exercise is an evidence-based treatment option that improves pain and disability outcomes in adults with osteoarthritis, but previous research has shown that adherence to prescribed exercise is low. Referral to physical therapy is common for people with OA with the standard of care including exercise prescription through paper handouts with brief instruction and static pictures. Such approaches do not incorporate known determinants of behavior change related to exercise adherence.

Recent technology products such as mobile applications (apps) for phones and tablets offer the potential to enhance communication between physical therapists and patients. The investigators aim to test a pragmatic intervention focused on supporting people with osteoarthritis to remain engaged with an exercise program. The specific aims of the project are to:

1. Compare the effectiveness of mobile app supported exercise prescription to usual care (paper exercise prescription) on exercise adherence among mid-life and older adults receiving similarly dosed physical therapy for lower extremity OA. The investigators will also examine secondary outcomes of exercise self-efficacy, physical function, stiffness, and pain.
2. Examine the feasibility and acceptability of mobile app supported exercise prescription through recruitment and retention rates, satisfaction with care ratings, and qualitative feedback.

ELIGIBILITY:
Inclusion Criteria:

1. Self-report of healthcare provider diagnosed osteoarthritis in the hips or knees
2. Ability to speak and read English
3. No diagnosis of serious mental illness
4. No diagnosis of serious or terminal illness (e.g., metastatic cancer, end stage renal failure)
5. Access to smartphone/tablet

Exclusion Criteria:

1. Cortisone injection to the joint with OA within the past 30 days
2. Undergoing physical therapy post-total joint replacement or in preparation for total joint replacement in the next 3 months
3. History of physical therapy for treatment of osteoarthritis in the past 6 months.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Exercise adherence | 0, 6, and 12 weeks
  Mean weekly exercise frequency over 6 and 12 weeks:0-21 with higher scores indicating more adherence.

SECONDARY OUTCOMES:
ShortMAC Physical Function Patient Reported Outcome MeasureRO | 0, 6 and 12 weeks
  12-item assessment of pain and function in people with osteoarthritis: 0-100 scale with higher scores for higher function and less pain
2 minute walk test | 0, 6 and 12 weeks
  Functional exercise capacity: Score is in meters/feet with higher distances indicating better exercise capacity
Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP) | 0, 6 and 12 weeks
  Pain measure: Scale range 0-100 with higher scores indicating worse pain
Timed Up and Go (TUG) + Dual Task | 0, 6 and 12 weeks
  Measure of physical function: Score is in seconds with higher scores indicating worse physical function
Dynamic Balance: Four square balance test | 0, 6 and 12 weeks
  Test of dynamic balance: Score is in seconds with lower scores indicating better dynamic balance
Self-efficacy for exercise (SEE) Scale | 0, 6, and 12 weeks
  Self-Efficacy for Exercise Scale: Score range 0-90 with higher score indicating higher self-efficacy for exercise

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Gell, PT, PhD, Principal Investigator — University of Vermont
Locations (1):
- Dee Physical Therapy, South Burlington, Vermont, United States